CLINICAL TRIAL: NCT06463119
Title: Registry of Vaccine Responses in Immune Compromised Patients
Acronym: REVAPI
Status: Recruiting | Type: Observational
Sponsor: Laure Pittet, MD-PhD (Other)
Responsible Party: Sponsor-Investigator, Laure Pittet, MD-PhD, Clinical Scientist, Pediatric Clinical Research Platform
Organization: Pediatric Clinical Research Platform (Other)
Other Study IDs: CCER 2024-00363
Record Dates: First submitted 2024-05-27; First posted 2024-06-17 (Actual); Last update posted 2024-11-07 (Actual); Status verified 2024-11

CONDITIONS: Immunosuppression
Keywords: Vaccine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples Without DNA — Provided sufficient funding, extra blood volume may be collected from a subset of participants for an in-dept evaluation of the immune response to vaccine, to evaluate vaccine-induced cellular response and memory cells, measured in the 1 to 3 months following vaccination (short-term response) and more than 9 months after vaccination (long-term response)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Immunocompromised patients: Priority will be given to patients with the following disease compromising their immune system:
  * Solid organ recipients
  * Hematopoietic stem cell transplant recipients
  * HIV
  * Dysimmune disorders
    * Inflammatory bowel disease
    * Rheumatologic disease
    * Neuro-immunological disease
    * Nephrotic syndrome
  * Primary immunodeficiency disorder
  * Pneumological disease requiring immunosuppression (e.g. bronchiolitis obliterans)
  * Oncological disease
  Interventions: Other: Collection of data in a registry

INTERVENTIONS:
Other: Collection of data in a registry — The aim of this observational project is to document the immunogenicity and reactogenicity of vaccines given to immunocompromised patients and collect it in a registry.

SUMMARY:
The aim of this project is to monitor, guide and document vaccination, vaccine responses, persistence of protection, vaccine efficacy and safety in immune compromised patients at various moment of their disease: right after the diagnosis, before the introduction of the immunosuppressive treatment, once the individual is under immunosuppressive treatment, or once immunosuppression is over.

DETAILED DESCRIPTION:
The aim of this project is to monitor, guide and document vaccination, vaccine responses, persistence of protection, vaccine efficacy and safety in immune compromised patients at various moment of their disease: right after the diagnosis, before the introduction of the immunosuppressive treatment, once the individual is under immunosuppressive treatment, or once immunosuppression is over. The project will not only help to optimise the vaccination status of the immunocompromised patients followed in our institution, but will enable to gather essential data on vaccine responses and the evolution of serology against vaccine-preventable diseases over time. The project will also collect essential data on vaccination with live-attenuated vaccines.

The University Hospitals of Geneva and the Centre of vaccinology of the University of Geneva are recognised worldwide for their expertise in vaccinology, particularly in immunocompromised patients. Unfortunately, the management of these patients is not yet standardised, and no data is collected, precluding its dissemination. The aim of this project is to enable to share our expertise on vaccination of immune compromised patients with other teams by standardizing our practice and creating a registry.

Although measles-mumps-rubella (MMR) and varicella-zoster virus (VZV) vaccination are recommended in selected immune compromised patients fulfilling strict safety criterion, these criteria are not standardised, and only few groups have reported on the immunogenicity and the safety of these vaccination. As a results, many healthcare providers are hesitant to administer the vaccines and call for standardized operating procedures for vaccination and follow-up that are adapted to each immunocompromised condition. In addition, there are no data on the patients' perceptions of these vaccinations.

Therefore, the objective of this project is to optimise the administration of vaccines to immunocompromised patients by providing tailored information and personalised follow-up. The project will evaluate what information the patients need before and after vaccination, and what kind of follow-up is the most appropriate for each condition. By providing a standardised clinical and serological follow-up, this project will also document the reactogenicity and the immunogenicity of vaccines, and identify whether they differ among the various immune compromised state. It will also identify in whom and for which vaccines, additional doses are required to reach protection, and in whom repeated doses are needed during follow-up to maintain protection throughout the years. The results of this project will help to improve the follow-up of immune compromised patients following vaccination, and provide tailored follow-up for each of the immune compromised condition.

ELIGIBILITY:
Inclusion Criteria:

1. Immune compromised patient or patient who will soon be immunocompromised
2. Informed consent as documented by signature

Exclusion Criteria:

1. Individual/parental inability to follow the procedures of the study, e.g. due to language problems, psychological disorders, known/suspected non-compliance, substance abuse, etc.
2. Plan to move out of the country or have prolong absence in the next 2 months

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Priority will be given to patients with the following disease compromising their immune system:
  * Solid organ recipients
  * Hematopoietic stem cell transplant recipients
  * HIV
  * Dysimmune disorders
    * Inflammatory bowel disease
    * Rheumatologic disease
    * Neuro-immunological disease
    * Nephrotic syndrome
  * Primary immunodeficiency disorder
  * Pneumological disease requiring immunosuppression (e.g. bronchiolitis obliterans)
  * Oncological disease
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2024-09-24 (Actual); Primary Completion 2029-04 (Estimated); Study Completion 2029-04 (Estimated)

PRIMARY OUTCOMES:
Number of dose of vaccine required to reach seroprotection | 2 months (window allowed: 1 to 3 months) after vaccination
  Number of doses of vaccines required to reach seroprotection, described by vaccine type and immunocompromised state

SECONDARY OUTCOMES:
Number of dose of vaccine required to maintain seroprotection | 5 years follow-up
  Number of doses of vaccines required to reach seroprotection, described by vaccine type and immunocompromised state
Immunogenicity of vaccine (vaccine responses) in immune compromised patients | 2 months (window allowed: 1 to 3 months) after vaccination
  Vaccine-induced seroprotection (defined as vaccine-specific immunoglobulin concentration above seroprotection cut-off) measured in the 1 to 3 months following vaccination. If funding is sufficient, vaccine-induced cellular response and memory cells will be quantified in a subgroup of participants. Correlation with clinical protection will be evaluated as well.
Persistence of vaccine-induced seroprotection in immune compromised patients | 5 years follow-up
  Persistence of vaccine-induced seroprotection (defined as vaccine-specific immunoglobulin concentration above seroprotection cut-off) measured more than 9 months after vaccination. There may be multiple measures per patients, as these are monitored regularly in immune compromised patients. If funding is sufficient, vaccine-induced functional antibodies, cellular responses and memory cells will be quantified in a subgroup of participants. Correlation with clinical protection will be evaluated as well.
Occurence of adverse event following vaccine administration in immune compromised patients | 0 to 42 days after vaccination
  Occurrence and severity of local and systemic reaction measured from day 0 to day 42 after vaccination
Patients' acceptability of the standardized follow-up | 5 years follow-up
  Evaluated through satisfaction questionnaire with open questions, qualitative research

CONTACTS AND LOCATIONS:
Overall Officials: Laure F Pittet, MD-PhD, Principal Investigator — University Hospitals of Geneva
Locations (1):
- University Hospitals of Geneva, Geneva, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided